CLINICAL TRIAL: NCT02317445
Title: Beijing Tiantan Hospital,Capital Medical University.
Brief Title: Relationship of Helicobacter Pylori Eradication Therapy and Long-term Outcome in Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Buxing Chen, Beijing Tiantan Hospital, Capital Medical University
Other Study IDs: HPERINACS
Record Dates: First submitted 2014-11-13; First posted 2014-12-16 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Acute Coronary Syndrome
Keywords: helicobacter pylori; eradication therapy; major adverse cardiac events; long-term outcome; To explore the significance of Hp eradication therapy in preventing major adverse cardiac events (MACE) and upper gastrointestinal bleeding (UGIB).
MeSH Terms: conditions — Acute Coronary Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Objective: To investigate the relationship between Helicobacter pylori (Hp) infection and the prognosis of acute coronary syndrome (ACS) in a Chinese population and to explore the significance of Hp eradication therapy in preventing major adverse cardiac events (MACE) and upper gastrointestinal bleeding (UGIB) in patients on dual antiplatelet treatment. Methods: To analyze 472 ACS patients with drug-eluting stent (DES) implantation from January 1, 2008 to December 31, 2010 in the department of cardiology at Beijing Mentougou District Hospital. Patients were divided into three groups: Group 1, the Hp-negative patients (Hp-); Group 2, the Hp-positive patients with eradication therapy (Hp+ Therapy); and Group 3, the Hp-positive patients without eradication therapy (Hp+ No Therapy). All patients took 13C urea breath test, high sensitive C-reactive protein (hs-CRP)，homocysteine (HCY) and other biochemical indicators. The investigators explored the correlations of Hp eradication therapy with MACE (including recurrent myocardial infarction, revascularization and death) and UGIB after 3 to 5 years of follow-up using survival analysis.

DETAILED DESCRIPTION:
This study is a single-center and random analysis. The consecutive hospitalized patients with ACS at Beijing Mentougou District Hospital from January 1, 2008 to December 31, 2010 were enrolled. Figure 1 is a flow diagram of the trial. There were 259 males (54.9%) and 213 females (45.1%) with an average age of 61.1 ± 11.0 years. Patient's history, physical examination, and laboratory results were recorded. All patients were divided into the Hp-negative group (Hp-, group 1.) and the Hp-positive group (Hp+). The Hp+ group were randomly divided into two groups: Group 2, the Hp+ with eradication therapy (Hp+ Therapy); and Group 3, the Hp+ without eradication therapy (Hp+No Therapy).

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed acute coronary syndrome according to the 2012 ESC guidlines.
* All the patients took dual antiplatelet therapy after implanting drug eluting stent (DES) during hospitalization and had no any digestive symptoms.

Exclusion Criteria:

* Subjects who had suffered gastrointestinal bleeding within one week.
* Subjects had a history of gastrectomy, cardiac insufficiency, thyroid dysfunction, and any ongoing infections were eliminated.
* Patients with the use of antibiotics, bismuth, or sucralfate within one month and without impanting DES because of ACS during hospitalization were also excluded.
* Those who had gastrointestinal symptoms, such as acid reflux, heartburn, nausea, vomiting, stomach ache and diarrhea, or had a confirmed peptic ulcer with Hp infection were excluded because these patients may be taken gastroenterology treatment.

Ages: 50 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a single-center and random analysis. The consecutive hospitalized patients with ACS at Beijing Mentougou District Hospital from January 1, 2008 to December 31, 2010 were enrolled. Figure 1 is a flow diagram of the trial. There were 259 males (54.9%) and 213 females (45.1%) with an average age of 61.1 ± 11.0 years. Patient's history, physical examination, and laboratory results were recorded. All patients were divided into the Hp-negative group (Hp-, group 1.) and the Hp-positive group (Hp+). The Hp+ group were randomly divided into two groups: Group 2, the Hp+ with eradication therapy (Hp+ Therapy); and Group 3, the Hp+ without eradication therapy (Hp+No Therapy).
Sampling Method: Non-Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the MACE among the three groups. | January 1, 2008 to December 31, 2013, up to 6 years
  The Hp+ without eradication therapy had more MACE than Hp-positive patients with eradication therapy

SECONDARY OUTCOMES:
Comparison of the upper gastrointestinal bleeding among the three groups. | January 1, 2008 to December 31, 2013, up to 6 years
  The Hp-infected patients without eradication therapy had more UGIB than Hp-positive patients with eradication therapy.

REFERENCES:
- [Result] Budzynski J, Klopocka M, Bujak R, Swiatkowski M, Pulkowski G, Sinkiewicz W. Autonomic nervous function in Helicobacter pylori-infected patients with atypical chest pain studied by analysis of heart rate variability. Eur J Gastroenterol Hepatol. 2004 May;16(5):451-7. doi: 10.1097/00042737-200405000-00003. PMID 15097036
- [Result] Fashner J, Gitu AC. Common Gastrointestinal Symptoms: dyspepsia and Helicobacter pylori. FP Essent. 2013 Oct;413:24-8. PMID 24124704
- [Result] Roesler BM, Rabelo-Goncalves EM, Zeitune JM. Virulence Factors of Helicobacter pylori: A Review. Clin Med Insights Gastroenterol. 2014 Mar 27;7:9-17. doi: 10.4137/CGast.S13760. eCollection 2014. PMID 24833944
- [Result] Ng FH, Wong SY, Lam KF, Chang CM, Lau YK, Chu WM, Wong BC. Gastrointestinal bleeding in patients receiving a combination of aspirin, clopidogrel, and enoxaparin in acute coronary syndrome. Am J Gastroenterol. 2008 Apr;103(4):865-71. doi: 10.1111/j.1572-0241.2007.01715.x. Epub 2008 Jan 2. PMID 18177451
- [Result] Lee SD. Notice of retraction of "The experience with Ritleng intubation system in patients with congenital nasolacrimal duct obstruction". J Chin Med Assoc 2004;67:344-8. J Chin Med Assoc. 2008 Jun;71(6):329. doi: 10.1016/S1726-4901(08)70133-3. No abstract available. PMID 18567567
- [Result] Rogha M, Nikvarz M, Pourmoghaddas Z, Shirneshan K, Dadkhah D, Pourmoghaddas M. Is helicobacter pylori infection a risk factor for coronary heart disease? ARYA Atheroscler. 2012 Spring;8(1):5-8. PMID 23056092
- [Result] Vafaeimanesh J, Hejazi SF, Damanpak V, Vahedian M, Sattari M, Seyyedmajidi M. Association of Helicobacter pylori infection with coronary artery disease: is Helicobacter pylori a risk factor? ScientificWorldJournal. 2014 Jan 16;2014:516354. doi: 10.1155/2014/516354. eCollection 2014. PMID 24574896
- [Result] Lee SY. Current progress toward eradicating Helicobacter pylori in East Asian countries: differences in the 2013 revised guidelines between China, Japan, and South Korea. World J Gastroenterol. 2014 Feb 14;20(6):1493-502. doi: 10.3748/wjg.v20.i6.1493. PMID 24587624
- [Result] Hamm CW, Bassand JP, Agewall S, Bax J, Boersma E, Bueno H, Caso P, Dudek D, Gielen S, Huber K, Ohman M, Petrie MC, Sonntag F, Uva MS, Storey RF, Wijns W, Zahger D; ESC Committee for Practice Guidelines. ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: The Task Force for the management of acute coronary syndromes (ACS) in patients presenting without persistent ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2011 Dec;32(23):2999-3054. doi: 10.1093/eurheartj/ehr236. Epub 2011 Aug 26. No abstract available. PMID 21873419
- [Result] Wright RS, Anderson JL, Adams CD, Bridges CR, Casey DE Jr, Ettinger SM, Fesmire FM, Ganiats TG, Jneid H, Lincoff AM, Peterson ED, Philippides GJ, Theroux P, Wenger NK, Zidar JP, Anderson JL, Adams CD, Antman EM, Bridges CR, Califf RM, Casey DE Jr, Chavey WE 2nd, Fesmire FM, Hochman JS, Levin TN, Lincoff AM, Peterson ED, Theroux P, Wenger NK, Wright RS. 2011 ACCF/AHA focused update of the Guidelines for the Management of Patients with Unstable Angina/Non-ST-Elevation Myocardial Infarction (updating the 2007 guideline): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines developed in collaboration with the American College of Emergency Physicians, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. J Am Coll Cardiol. 2011 May 10;57(19):1920-59. doi: 10.1016/j.jacc.2011.02.009. Epub 2011 Mar 28. No abstract available. PMID 21450428